CLINICAL TRIAL: NCT03084107
Title: LES_Cloud - Advanced Eldercare Technology and Creative Space
Brief Title: Eldercare Technology in a Silver Culture Village
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Alice May-Kuen Wong, Attending Physician, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 100-1075B
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Elderly
Keywords: Elder care; Active aging; Intelligent Care Facilities for Elders
MeSH Terms: interventions — Surveys and Questionnaires

ARMS (1):
- Questionnaire (Experimental): technology acceptance model (TAM) questionnaire
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The elderly participated in the application of smart devices and requested to complete technology acceptance model (TAM) questionnaires for these devices.

SUMMARY:
The aim of this project is to create ten smart devices that involve combining an interactive art environment with IC technology, arts and health administration. Investigators invited the elderly residents of Chang Gung Health and Culture Village to participate in the application of these devices, and participants were also requested to complete a technology acceptance model (TAM) questionnaire for these smart devices.

DETAILED DESCRIPTION:
According to statistics in Taiwan, by 2050, one-third population of Taiwan citizens will be over 65 years old. By the definition in World Health Organization, "Active aging" is the process of optimizing opportunities for health, participation and security in order to enhance the quality of life as people age. Active aging aims to extend healthy life expectancy and quality of life for all people as they age.

Chang Gung Health and Culture Village is one of the largest and most experienced aged care and retirement living providers in Taiwan.In this project, for promoting the successful aging of elderly residents, investigators will integrate health management systems and wireless sensor networks, physiological telemetry, learning and exercise behavior in Chang Gung Health and Culture Village. The investigators expect to build a Intelligent Care Facilities space for Elders base on exercise and rehabilitation with ten smart devices that involve combining an interactive art environment with computer science technology, multimedia applications and health administration in three years. Investigators invited the elderly residents to participate in the application of these devices, thereby increasing participants' physical activity and improving the physiological conditions. Participants were also requested to complete a technology acceptance model (TAM) questionnaire for these smart devices.

With respect to old age, long-term care is the human rights. How to provide an excellent eldercare to the elder people is a challenge. "Elder care", "Technology", "Art", "Medicine", a team of interdisciplinary experts is required to achieve this goal. The products of this study will promote an excellent elder care, in the setting of their choice by offering older people the information, services and support needed to make choices which enhance health, well-being and independence. In addition to analyze the acceptance model of intelligent care facilities for elders, the investigators expect the experience can help academic and industrial circles to research and develop care facilities for elders in the future.

ELIGIBILITY:
Inclusion Criteria:

* elderly who lived in the Chang Gung Health and Culture Village

Exclusion Criteria:

* inability to complete questionnaires

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-08-01; Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
TAM Questionnaire | 3 years
  The Design Quality and Interface positively raised Awareness of Fun for the elderly participants in these smart devices, and the Perceived Usefulness positively affects the participants' willingness to use the devices.

CONTACTS AND LOCATIONS:
Overall Officials: Alice MK Wong, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan